CLINICAL TRIAL: NCT00574483
Title: An Open-label, Fixed-dose, Clinical Study of Quinacrine Safety and Efficacy in the Treatment of Advanced Renal Cell Carcinoma
Brief Title: Treatment of Advanced Renal Cell Carcinoma With Quinacrine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: reevaluation of compound development
Sponsor: Cleveland BioLabs (Industry)
Responsible Party: John H. Gordon, Cleveland BioLabs, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBL-DD-07-C-H-2002
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2008-01

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Quinacrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Unblinded treatment arm
  Interventions: Drug: quinacrine

INTERVENTIONS:
Drug: quinacrine — 100 mg day
  Other Names: CBLC102

SUMMARY:
The overall response to standard therapies and to the newer antiangiogenesis therapies is not curative, and treatment-associated toxicities may be severe. Therefore, continued evaluation of therapies, with different mechanisms of action, is needed for patients with metastatic RCC.

DETAILED DESCRIPTION:
Approximately 31,000 new cases of renal cell carcinoma (RCC) occur each year in the United States, with a death rate of about 11,600 annually. Many patients present with advanced or unresectable disease, and up to 30% of patients who are treated with nephrectomy will relapse. The 5 year survival rate for metastatic renal RCC is estimated at < 10%. Surgical resection of discernible disease is the only potentially curative treatment. No significant improvement in survival has been demonstrated for patients with metastatic RCC who have been treated with systemic hormonal, chemotherapeutic, and radiation therapy. Interferon alpha has about a 15% objective response rate in appropriately selected patients. Administration of interleukin 2 (IL 2) has shown a similar response rate; however, approximately 5% of highly selected patients had durable complete remissions.

Recent studies demonstrated that RCC cells harbor abnormalities of the von Hippel-Lindau (VHL) gene, playing a key role in the stimulation of angiogenesis by vascular endothelial growth factor (VEGF) in this highly vascularized tumor. The novel agents sunitinib (Sutent) and sorafenib (Nexavar) are approved by the US Food and Drug Administration (FDA) for the treatment of advanced RCC, and both bevacizumab (Avastin) and temsirolimus have shown significant activity in treatment-naïve patients. Prolonged progression-free survival has been reported with sorafenib and sunitinib in randomized, controlled phase 2 and 3 studies, and improved survival has been reported with temsirolimus in poor-risk patients in a phase 3 randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed RCC with clear cell predominance.
* Subjects must provide written informed .
* Subjects must be at least 18 years old.
* Subjects must have at least 1 measurable lesion.
* Subjects must have metastatic, locally advanced or unresectable RCC.
* Subjects must have received ≥ 1 prior systemic regimen for RCC.
* All prior cancer therapy, including radiation, surgery, and systemic (hormonal, chemotherapeutic, and immunotherapeutic) therapy, must be completed at least 4 weeks before the baseline visit.
* Subjects must be capable of adhering to the study visit schedule and other protocol requirements.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Subjects must have:

  1. Absolute neutrophil count (ANC)> 1,500/uL
  2. Hemoglobin > 10.0 g/dL
  3. Platelets ≥ 100,000/uL
  4. Serum creatinine < 2.0 mg/dL
* Subjects must have adequate hepatic function, as defined by a bilirubin level of ≤ 1.5 times the upper limit of the normal range (ULN) and an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level of ≤ 3 times the ULN (or ≤ 5 times the ULN if liver metastases are present).
* Women of childbearing potential must have a negative serum pregnancy test at the screening visit and throughout the study.
* Sexually active women and men must agree to use a medically acceptable form of contraception.

Exclusion Criteria:

* Subjects who have a history of any malignancy (other than excised basal cell carcinoma or cervical intraepithelial neoplasia) within the 5 years of baseline visit.
* Subjects who have received any anticancer agents, treatment (chemotherapy, targeted agents, radiation, hormones), or investigational agents within 30 days of the baseline visit.
* Subjects who have untreated brain metastases.
* Subjects who have a history of hypersensitivity reaction to quinacrine or other acridine derivatives (e.g. Cognex).
* Subjects who have any clinically significant hematological, endocrine, cardiovascular (including any rhythm disorder), renal, hepatic, gastrointestinal (GI), or neurological disease (including any history of seizure).
* Subjects who have a history of porphyria or psoriasis.
* Subjects who have documented glucose-6-phosphate dehydrogenase deficiency.
* Subjects who have a history of noninfectious (toxic, autoimmune) hepatitis.
* Subjects who have a history of schizophrenia, bipolar disorder, or any psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects who have a history of dermatitis as an allergic/toxic reaction to any medication.
* Subjects who have any grade 2 sensory neuropathy.
* Subjects who have a QTcF (Fredericia) of > 450 msec.
* Subjects who have New York Heart Association (NYHA) class 3 or 4 heart failure.
* Subjects who had a myocardial infarction or acute coronary syndrome within 6 months of the baseline visit.
* Subjects who require anti-arrhythmic treatment with amiodarone or any drug with a quinidine-like effect on the heart or who have history of a malignant ventricular arrhythmia unless they have a functioning Automatic Implantable Cardio-Defibrillator (AICD) implanted.
* Subjects who are immunocompromised, including those known to be human immunodeficiency virus (HIV) positive, hepatitis B positive, or hepatitis C positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Estimated); Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 6 months

SECONDARY OUTCOMES:
Time to tumor progression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John H Gordon, PhD, Study Director — Cleveland BioLabs
Locations (2):
- United States (2):
  - Community Care Physicians, Albany, New York
  - ClinWorks Cancer Research Center, Charlotte, North Carolina